CLINICAL TRIAL: NCT05443204
Title: Evaluation of Glycemic Control by Flash Monitoring of Glucose (MFG) in Malnourished Patients With Type 2 Diabetes and Oral Supplements: Standard Formula vs Specific Formula for Diabetes
Brief Title: Evaluation of Glycemic Control by Flash Monitoring of Glucose (MFG) in Malnourished Patients With Type 2 Diabetes
Acronym: MFG-SNO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MFG SNO
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Type 2; Malnutrition
Keywords: Diabetes type 2; Malnutrition; MFG
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Malnutrition

STUDY DESIGN:
Intervention Model Description: Patients will be assigned in a 1:1 ratio
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Formula (Fortimel) (Experimental): Fats 35% total caloric volume (VCT) Carbohydrates: 49% del VCT Proteins: 16% del VCT Density: 1.5 kcal/ ml
  Interventions: Other: Fortimel energy
- Specific formula for diabetes (Nutrision Advanced) (Experimental): Fats: 46% del VCT (60% monounsaturated fatty acids) Carbohydrates: 31% del VCT Proteins: 21% del VFiber: 2% VCT (80% soluble y 20% insoluble) Density: 1.5kcal/ml
  Interventions: Other: Nutrision Advanced Diason Energy HP

INTERVENTIONS:
Other: Fortimel energy — Standard nutritional oral supplement
  Arms: Standard Formula (Fortimel)
Other: Nutrision Advanced Diason Energy HP — Specifc nutritional oral supplement in diabetics patients
  Arms: Specific formula for diabetes (Nutrision Advanced)

SUMMARY:
Evaluation of Glycemic Control by Flash Monitoring of Glucose (MFG) in Malnourished Patients With Type 2 Diabetes (MFG SNO)

DETAILED DESCRIPTION:
In people with malnutrition and diabetes who require oral supplementation, there is no evidence clear when choosing a specific supplement for diabetes or a standard supplement. To date, there are no studies evaluating flash glucose monitoring in people with DM2 with supplements, nor studies comparing formulas specific for diabetes with standard formulas. Patients with type 2 diabetes, malnutrition and requiring oral nutritional supplements for 3 months will be included in the study.

A standard supplement (minimum 2 per day) will be prescribed for 2 weeks, an installation of the MFG system indicating that the scans are performed at start up, at the time and two hours after taking the oral supplement at home, as it doesn't happen anymore 8 hours without scanning to avoid losing information. After 14 days participants will go to consultation to download MFG data, assess acute response after taking of the supplement in the presence of health personnel (every 15 minutes for 4 hours). Investigators will change the sensor and nutritional supplement to a specific diabetes formula, after 14 days participants will come for MFG data download and to assess acute response after taking the supplement in the presence of healthcare personnel.

The results of the study will allow us to carry out a more appropriate treatment in this profile of patients, which is increasingly prevalent in our consultations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DM2 under follow-up by the Clinical Nutrition and Dietetics Unit (UNCYD) who present malnutrition or are at risk of malnutrition and require oral nutritional supplements, for a minimum estimated period of 3 months.

Exclusion Criteria:

* Patients with DM1, steroid diabetes, pancreatic diabetes, DM2 treated with rapid insulin, glomerular filtration rate less than 30 mL/min/1.73m2, intolerance to the product, gastrectomy or gastroparesis.
* Patients who do not sign the consent informed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
MFG discharge - mean interstitial glucose | During 14 days after taking the supplement
  Interstitial glucose measured in mg/dl
MFG discharge - hyperglycaemia | During 14 days after taking the supplement
  hyperglycaemia measured in mg/dl
MFG discharge - hypoglycaemia | During 14 days after taking the supplement
  hypoglycaemia measured in mg/dl
MFG discharge - GMI | During 14 days after taking the supplement
  Measured in number of scans per day
MFG discharge - hypoglycaemic events | During 14 days after taking the supplement
  Measured in number and duration per day

SECONDARY OUTCOMES:
Postprandial glucose intersticial monitoringdiabetes specific supplement | During the 4 hours after taking standard formula and the one specific for diabetes
  Glucose intersticial measured in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Olveira Fuster, MD, PhD., Principal Investigator — Hospital Regional Universitario de Málaga - FIMABIS
Locations (1):
- Hospital Regional Universitario de Málaga, Málaga, Spain